CLINICAL TRIAL: NCT02911064
Title: Assessment of Expectations Regarding Mobility and Self-Care Between Physiatrists and Oncology Patients
Brief Title: Expectations Regarding Mobility and Self-Care
Status: Active, not recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-0550; NCI-2018-01760 (Other: NCI-CTRP-Clinical Trial Reporting Registry)
Record Dates: First submitted 2016-09-16; First posted 2016-09-22 (Estimated); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Benign Neoplasms; Malignant Neoplasms of Independent (Primary) Multiple Sites
Keywords: Questionnaires; Surveys; Benign neoplasms; Malignant neoplasms of independent (primary) multiple sites; Inpatient rehabilitation therapy
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assessment Questionnaires: Questionnaires completed before and after inpatient rehabilitation. Questionnaires ask about daily living activity performance, expectation of how well daily living activities will be performed after completion of inpatient rehabilitation, symptoms experienced in the past 24 hours, and physical, functional, social, and emotional well-being.
  Interventions: Behavioral: Questionnaires

INTERVENTIONS:
Behavioral: Questionnaires — Questionnaires completed before and after inpatient rehabilitation. Questionnaires ask about daily living activity performance, expectation of how well daily living activities will be performed after completion of inpatient rehabilitation, symptoms experienced in the past 24 hours, and physical, functional, social, and emotional well-being. These questionnaires should take about 15 minutes total to complete.
  Other Names: Surveys

SUMMARY:
The goal of this research study is to learn if there is a difference between your expectations of how well you will perform daily living activities after short-term inpatient rehabilitation and the doctor's expectations of how well you will perform daily living activities.

DETAILED DESCRIPTION:
If you agree to take part in this study, you will complete questionnaires before your inpatient rehabilitation and after you complete inpatient rehabilitation. The questionnaires will ask about how well you currently perform daily living activities, your expectation of how well you will perform daily living activities after you complete inpatient rehabilitation, your symptoms in the past 24 hours, and your physical, functional, social, and emotional well-being. These questionnaires should take about 15 minutes total to complete.

Information from your medical record (such as your age, gender, religion, cancer diagnosis, stage of cancer, and so on) will be collected.

Length of Study:

You participation on this study will be over after you complete the questionnaires.

This is an investigational study.

Up to 111 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are willing and able to give written informed consent and to comply with all of the study visits and surveys
2. Patients with any type of cancer admitted on the acute inpatient rehabilitation unit who can tolerate 3 hours of rehabilitation therapies per day
3. Patients 18 years and older
4. Patients must be able to understand, read, write, and speak English.

Exclusion Criteria:

1. Patients who have delirium, severe symptom distress, or cognitive impairment.
2. Patients who return to primary service prior to discharge from the acute inpatient rehabilitation unit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants scheduled to receive inpatient rehabilitation therapy at University of Texas MD Anderson Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 133 (Actual)
Dates: Start 2016-11-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of Participant and Physiatry Practitioner Expectations of Mobility and Activities of Daily Living After Acute Inpatient Rehabilitation Using Barthel Index | 3 days
Assessment of Participant and Physiatry Practitioner Expectations of Mobility and Activities of Daily Living After Acute Inpatient Rehabilitation Using Eastern Cooperative Oncology Group (ECOG) Performance Status Scales | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Ekta Gupta, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org